CLINICAL TRIAL: NCT00559806
Title: The Effect of Aging and Immobilisation on Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: KF01-322606
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: Healthy
Keywords: immobilisation; aging; resistance training; atrophy; The effect of immobilisation in elderly compared to young individuals
MeSH Terms: conditions — Atrophy | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 9 healthy elderly males
  Interventions: Other: 2 weeks of unilateral immobilisation and 4 weeks of resistance training
- 2 (Experimental): 11 healthy young males
  Interventions: Other: 2 weeks of unilateral immobilisation and 4 weeks of resistance training

INTERVENTIONS:
Other: 2 weeks of unilateral immobilisation and 4 weeks of resistance training — 2 weeks of whole leg casting (side randomized)followed by 4 weeks of unilateral resistance training. The non-imm side served as a within-subject control
  Arms: 1
Other: 2 weeks of unilateral immobilisation and 4 weeks of resistance training — 2 weeks of unilateral whole leg casting (side randomized)followed by 4 weeks of unilateral resistance training. The non-imm side served as a within-subject control
  Arms: 2

SUMMARY:
The debilitating effects of immobilisation on muscle strength and size in young individuals are well documented. Moreover, sarcopenia has long been recognized as a major cause of muscle strength loss in old age, however, changes in muscle mass and architecture with immobilisation in the elderly has not previously been investigated. This is contrasted by the fact that the elderly population more often undergoes periods of immobilization and disuse not only due to joint pain but also due to a higher degree of co morbidity and hospitalisation.The purpose of the present study was to compare the effect of a 2 week period of unilateral immobilisation on the physiological muscle cross sectional area, maximal isometric muscle strength, specific force, muscle fascicle length and muscle fibre pennation angle in young and old healthy men.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy males (age 20-30 yrs)or old healthy males (age 60-80 yrs)

Exclusion Criteria:

* Musculoskeletal disorder
* Diabetes
* Cardiovascular disease
* Neurological diseases; or
* Cognitive disorders

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
muscle cross sectional area, maximal isometric muscle strength, specific force, muscle fascicle length and muscle fibre pennation | 2 weeks of immobilisation and 4 weeks of resistance training

SECONDARY OUTCOMES:
single muscle fiber area, expression of myostatin and IGF-1 (RNA), changes in satellite activation and number | 2 weeks of imm and 4 weeks of resistance training

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Suetta, MD, PhD, Principal Investigator — Institute of Sports Medicine Copenhagen, Bispebjerg Hospital
Locations (1):
- Institute of Sports Medicine, Bispebjerg Hospital, Copenhagen, Denmark